CLINICAL TRIAL: NCT06911684
Title: Short-Term Radiotherapy Combined With Iparomlimab and Tuvonralimab (QL1706), Regorafenib, and CAPOX Neoadjuvant Therapy for Locally Advanced Rectal Cancer：A Multicenter, Prospective, Randomized, Phase II Clinical Trial
Brief Title: Radiotherapy Plus Iparomlimab and Tuvonralimab (QL1706), Regorafenib, and CAPOX as Neoadjuvant Therapy for pMMR/MSS LARC.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Director of the Department of Colorectal Surgery, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-149
Record Dates: First submitted 2025-03-15; First posted 2025-04-04 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer Patients
Keywords: Rectal Cancer; Neoadjuvant Therapy; pMMR/MSS; immunotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A patients received two cycles of QL1706, regorafenib, and CAPOX induction therapy, followed by sequential short-course radiotherapy, and then continued with four cycles of QL1706, regorafenib, and CAPOX consolidation therapy.
  Interventions: Combination Product: lparomlimab and Tuvonralimab Injection and regorafenib and CPAOX and short-course radiotherapy
- Group B (Experimental): Group B patients received short-course radiotherapy followed by six cycles of QL1706, regorafenib, and CAPOX consolidation therapy.
  Interventions: Combination Product: lparomlimab and Tuvonralimab Injection and regorafenib and CPAOX and short-course radiotherapy

INTERVENTIONS:
Combination Product: lparomlimab and Tuvonralimab Injection and regorafenib and CPAOX and short-course radiotherapy — Group A patients received two cycles of QL1706, regorafenib, and CAPOX induction therapy, followed by sequential short-course radiotherapy, and then continued with four cycles of QL1706, regorafenib, and CAPOX consolidation therapy.
  lparomlimab and Tuvonralimab Injection(QL1706): 5 mg/kg, intravenous (IV), on Day 1, every 3 weeks (q3w) during the neoadjuvant treatment phase.
  Regorafenib:80 mg, oral (PO), once daily (qd), Days 1-14, every 3 weeks (q3w) during the neoadjuvant treatment phase.
  CAPOX: Oxaliplatin( 130 mg/m², IV over 2 hours, Day 1, every 3 weeks (q3w))+ Capecitabine( 1000 mg/m², PO, twice daily (bid), Days 1-14, every 3 weeks (q3w)).
  Short-course radiotherapy:The total dosage was 25Gy consisted of 5 fractions of 5 Gy to clinical target volume without a boost dose.
  Arms: Group A
Combination Product: lparomlimab and Tuvonralimab Injection and regorafenib and CPAOX and short-course radiotherapy — Group B patients received short-course radiotherapy followed by six cycles of QL1706, regorafenib, and CAPOX consolidation therapy.
  lparomlimab and Tuvonralimab Injection(QL1706): 5 mg/kg, intravenous (IV), on Day 1, every 3 weeks (q3w) during the neoadjuvant treatment phase. Regorafenib:80 mg, oral (PO), once daily (qd), Days 1-14, every 3 weeks (q3w) during the neoadjuvant treatment phase. CAPOX: Oxaliplatin( 130 mg/m², IV over 2 hours, Day 1, every 3 weeks (q3w))+ Capecitabine( 1000 mg/m², PO, twice daily (bid), Days 1-14, every 3 weeks (q3w)). Short-course radiotherapy:The total dosage was 25Gy consisted of 5 fractions of 5 Gy to clinical target volume without a boost dose.
  Arms: Group B

SUMMARY:
This study is a multicenter, prospective, randomized, double-arm, Phase II clinical trial designed to evaluate the efficacy of short-term radiotherapy combined with Iparomlimab and Tuvonralimab (QL1706), Regorafenib, and CAPOX as neoadjuvant therapy for locally advanced rectal cancer. Additionally, the study seeks to explore the relationship between biomarkers in blood, urine, feces, and tumor tissue and treatment efficacy.

Eligible participants (pMMR/MSS locally advanced rectal cancer) were randomly assigned in a 1:1 ratio to two groups, with randomization stratified by MRF (+ vs. -).

Participants will:

* Group A patients received two cycles of QL1706, regorafenib, and CAPOX induction therapy, followed by sequential short-course radiotherapy, and then continued with four cycles of QL1706, regorafenib, and CAPOX consolidation therapy.
* Group B patients received short-course radiotherapy followed by six cycles of QL1706, regorafenib, and CAPOX consolidation therapy.

After two cycles of neoadjuvant therapy in Group A and six cycles in Group B, efficacy was evaluated and decisions regarding surgery or watchful waiting were made based on efficacy.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common malignancy worldwide. The standard treatment for locally advanced rectal cancer (LARC) includes neoadjuvant chemoradiotherapy, total mesorectal excision (TME), and postoperative adjuvant chemotherapy. However, distant metastasis and postoperative complications remain major challenges. Total neoadjuvant therapy (TNT), by advancing adjuvant chemotherapy to the neoadjuvant phase, has significantly improved patient compliance and tumor response rates. The MSKCC study demonstrated a tumor response rate of up to 90% under the TNT regimen, with 30% of patients achieving pathological or clinical complete response (pCR or cCR). The TIMING trial further confirmed that TNT significantly increased the pCR rate without increasing side effects or surgical complications.

Immunotherapy has shown significant efficacy in dMMR/MSI-H CRC. The NICHE study demonstrated that dual immunotherapy achieved 100% pathological response in dMMR colorectal cancer patients. However, pMMR/MSS CRC is not sensitive to immunotherapy, but some patients may still benefit from combined anti-angiogenesis agents (such as regorafenib) or CTLA-4 antibodies. The REGONIVO study showed an objective response rate (ORR) of 36.0% in pMMR/MSS CRC patients, while the RIN study further increased the ORR to 27.6%.

Radiotherapy combined with immunotherapy has emerged as a new treatment modality for LARC. The UNION study found that short-term radiotherapy followed by sequential PD-1 antibody and CAPOX chemotherapy increased the pCR rate to 39.8%. The TORCH study explored the effectiveness of short-term radiotherapy combined with PD-1 antibody and CAPOX chemotherapy, achieving a CR rate of over 50%. The REGINA study went further, using short-term radiotherapy combined with regorafenib and nivolumab, achieving a CR rate of 44.4%.

Iparomlimab and Tuvonralimab (QL1706) is a bispecific antibody targeting PD-1 and CTLA-4, enhancing T cell activation and anti-tumor response through synergistic effects. In September 2024, QL1706 was approved for the treatment of recurrent or metastatic cervical cancer. Based on existing studies, short-term radiotherapy combined with immunotherapy (PD-1 antibody, CTLA-4 antibody), regorafenib, and CAPOX chemotherapy may significantly improve efficacy in pMMR/MSS LARC patients, warranting further exploration of its safety and effectiveness.

Eligible participants (pMMR/MSS locally advanced rectal cancer) were randomly assigned in a 1:1 ratio to two groups, with randomization stratified by MRF (+ vs. -). Group A patients received two cycles of QL1706, regorafenib, and CAPOX induction therapy, followed by sequential short-course radiotherapy, and then continued with four cycles of QL1706, regorafenib, and CAPOX consolidation therapy. Group B patients received short-course radiotherapy followed by six cycles of QL1706, regorafenib, and CAPOX consolidation therapy. After two cycles of neoadjuvant therapy in Group A and six cycles in Group B, efficacy was evaluated and decisions regarding surgery or watchful waiting were made based on efficacy. Postoperative need for adjuvant therapy was determined by the investigator.

Efficacy assessment: Patients achieving clinical complete response (cCR) could undergo a watch-and-wait strategy; patients with near cCR could undergo transanal local excision; patients with partial response (PR) or stable disease (SD) would undergo radical surgery. The need for postoperative adjuvant therapy was determined by the investigator. Patients with local progressive disease (PD) or distant metastasis were treated according to current guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years.
2. Pathology: Histologically confirmed rectal adenocarcinoma, with the lower tumor edge ≤12 cm from the anal verge.
3. Initial Clinical Stage: cT3-4aN0M0 or cT1-4aN+M0, regardless of MRF, EMVI, or LLNM status.

   Preoperative staging methods: chest and abdominal CT, pelvic MRI, endoscopic ultrasound (EUS), or transrectal ultrasonography.
4. pMMR/MSS Status: pMMR confirmed by immunohistochemistry (IHC) at the study center's pathology department, or MSS/MSI-L confirmed by PCR or NGS.
5. ECOG Performance Status: 0-1.
6. Informed Consent: Voluntarily agrees to participate and signs the informed consent form.
7. No Prior Treatment: No previous therapy targeting rectal adenocarcinoma, including radiotherapy, chemotherapy, or surgery.
8. Planned Surgery: Surgery is planned upon completion of neoadjuvant therapy.
9. Expected Survival: ≥6 months.
10. Adequate Organ and Bone Marrow Function, meeting all of the following (with no blood products, growth factors, or other hematopoietic-supportive medications used within 14 days before first administration):

    Hematology:

    Absolute neutrophil count (ANC) ≥1.5 × 10^9/L Platelet count ≥100 × 10^9/L Hemoglobin ≥90 g/L

    Serum Biochemistry:

    Serum albumin ≥30 g/L Total bilirubin ≤1.5 × ULN ALT ≤2.5 × ULN, AST ≤2.5 × ULN Alkaline phosphatase (ALP) ≤2.5 × ULN

    Serum creatinine ≤1.5 × ULN, or creatinine clearance (CrCl) ≥50 mL/min, calculated by the Cockcroft-Gault formula:
11. Contraception:

    Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the first study dose, and must use effective contraception (e.g., intrauterine device, oral contraceptive, or barrier method) during the study and for at least 120 days after the final dose.

    Male participants with partners of childbearing potential must be surgically sterile or must agree to use effective contraception during the study and for 120 days after the final dose.
12. Compliance and Follow-up: Demonstrates good compliance and agrees to attend follow-up visits.
13. Biological Samples: Agrees to provide blood, urine, stool, and tumor tissue samples.

Exclusion Criteria:

1. Active Autoimmune Disease: Any active autoimmune disease requiring systemic treatment (i.e., disease-modifying medications, corticosteroids, or immunosuppressive agents) within 2 years prior to enrollment (e.g., myasthenia gravis, systemic lupus erythematosus, interstitial pneumonitis, uveitis, ulcerative colitis, autoimmune hepatitis, hypophysitis, systemic vasculitis, nephritis, hyperthyroidism, hypothyroidism, mixed connective tissue disease).

   Exceptions: vitiligo, or childhood asthma that has fully resolved in adulthood without therapy.

   Asthma requiring bronchodilator therapy is ineligible. Physiologic replacement therapy (e.g., thyroid hormone, insulin, or low-dose steroids for adrenal/pituitary insufficiency) is not considered systemic treatment.
2. Concurrent Systemic Therapy: Use of systemic corticosteroids (≥10 mg/day of prednisone or equivalent) or other immunosuppressants (e.g., cyclosporine, cyclophosphamide, azathioprine, methotrexate, thalidomide) within 14 days before the first dose, or use of immunostimulants (e.g., interferon, interleukin-2) within 4 weeks before the first dose.
3. Live Vaccines: Receipt of a live or attenuated live vaccine within 30 days before the first dose or potentially during the study period.
4. Antibiotic Use: Administration of broad-spectrum antibiotics by any route within 30 days prior to the first dose.
5. Previous Anticancer Therapies: Any prior antitumor treatments (radiotherapy, chemotherapy, surgery [excluding biopsy], PD-1/CTLA-4 dual immunotherapy, regorafenib, or other tyrosine kinase inhibitors).
6. Unresectable Factors: Tumors deemed unresectable or participants with surgical contraindications, or who refuse surgery.
7. Immunodeficiency: HIV infection, any other acquired or congenital immunodeficiency disorder, or a history of organ or allogeneic bone marrow transplantation (excluding corneal transplantation).
8. Hepatitis B/C Co-infection:

   HBsAg-positive and/or HBcAb-positive with HBV DNA >10^4 copies/mL (≈2000 IU/mL).

   Anti-HCV antibody-positive with HCV-RNA >10^3 copies/mL. Patients positive for both HBsAg and HCV-RNA are excluded.
9. Other Malignancies: Any other malignancies within the past 5 years or concurrent malignancies, except for treated basal cell carcinoma of the skin or carcinoma in situ of the cervix.
10. Uncontrolled Effusions: Uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage.
11. Severe Pulmonary Conditions: Known active pulmonary tuberculosis, radiation pneumonitis, drug-induced pneumonitis, or other severe pulmonary diseases/impairments.
12. Renal Failure: Renal failure requiring hemodialysis or peritoneal dialysis.
13. Active Infection or Fever: Active infection, unexplained fever ≥38.5°C within 7 days prior to study treatment, or baseline WBC count >15 × 10^9/L.
14. Cardiac Conditions: Poorly controlled or clinically significant cardiac conditions, including:

    NYHA Class II or higher heart failure, LVEF <50% Unstable angina Myocardial infarction within 1 year prior to randomization Clinically significant arrhythmias requiring treatment or intervention QTc >450 ms (men), or QTc >470 ms (women)
15. Hypertension: Poorly controlled (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg) despite antihypertensive therapy, or a history of hypertensive crisis/encephalopathy.
16. Recent Thrombosis: Arterial or venous thrombosis within 6 months prior to enrollment (e.g., stroke, transient ischemic attack, cerebral hemorrhage, cerebral infarction, deep vein thrombosis, pulmonary embolism).
17. Coagulopathy: Known hereditary or acquired bleeding/thrombotic disorders (e.g., hemophilia, coagulopathy).
18. Significant Bleeding: Evidence or history of bleeding. Any Grade ≥3 hemorrhage within 4 weeks prior to study treatment (per CTCAE v5.0).
19. Vascular Invasion: Tumor invasion of major blood vessels or a high likelihood thereof during the study, potentially leading to life-threatening bleeding as judged by imaging.
20. Wounds or Ulcers: Severe, unhealed or dehiscent wounds, active ulcers, or untreated fractures.
21. Major Vascular Disease: Major vascular disorders within 6 months prior to study treatment (e.g., requiring surgical repair for an aneurysm or recent peripheral arterial thrombosis).
22. Major Surgery: Major surgery (other than diagnostic) within 4 weeks prior to study treatment, or planned major surgery during the study period (excluding the planned study-related procedure).
23. Abdominal Fistula, Perforation, or Abscess: Such events within 6 months prior to study treatment.
24. Long-Term NSAIDs or Anticoagulants: Need for long-term or high-dose NSAIDs (≥325 mg aspirin) or anticoagulant therapy.
25. Known Drug Allergy: Suspected or known allergy to any study drug or its components relevant to this trial.
26. Monoclonal Antibody Hypersensitivity: History of severe hypersensitivity reactions to any monoclonal antibody, or known hypersensitivity/allergy to QL1706, regorafenib, oxaliplatin, capecitabine, or any of their components.
27. Difficulty Swallowing: Inability or difficulty swallowing oral study drugs.
28. Pregnant or Breastfeeding: Women who are pregnant or lactating.
29. Other Factors: Any other factors that may affect study outcomes or lead to premature termination, including a history of alcohol or drug abuse, severe diseases (including psychiatric disorders) requiring combination treatment, significant laboratory abnormalities, or family/social circumstances that, in the investigator's judgment, compromise patient safety or study integrity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) | 1 year
  Complete response: Pathological complete response and clinical complete response

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year
  The proportion of patients achieving a complete response (CR) or partial response (PR), evaluated according to RECIST v1.1.
Major Pathological Response (MPR) | 1 year
  The proportion of patients whose primary tumor shows ≤10% residual tumor cells on pathology.
Tumor Regression Grade (TRG) | 1 year
  Assessed based on the 8th edition of the AJCC staging system to grade the extent of tumor regression
R0 Resection Rate | 1 year
  The proportion of surgical patients who achieve an R0 resection. R0 resection: All gross disease has been removed, and microscopic examination reveals all surgical margins free of tumor.
Organ Preservation Rate (OPR) | 1 year
  The 1-year organ preservation rate is the percentage of patients attaining a complete clinical response (cCR) or near-complete clinical response (near-cCR) following neoadjuvant therapy, who then proceeded with non-surgical management or local excision, was monitored under a Watch & Wait strategy or for 1 year post-local resection without undergoing radical surgery.
Event-free survival (EFS) | 2 years
  EFS is defined as the time from randomization to the earliest occurrence of any of the following events:
  Tumor progression by imaging according to RECIST 1.1, Tumor recurrence (local or distant), confirmed by imaging or biopsy, for patients with no residual tumor after surgery, Death from any cause. Note: A second primary malignancy is not considered an EFS event.
Overall survival (OS) | 5 years
  The time interval between the date of randomization to the date of death. If the patient has been alive, the time until the last follow-up is taken as the overall survival period.
Incidence of adverse events | up to 30 days after last treatment
  Assessed by Common Terminology Criteria for Adverse Events version 4.0. The overall adverse event rates and the immune-related adverse event rates will be compared between treatment arms using Chi-square test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Ding M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Dept. of Colorectal Surgery, Sun Yat-sen University Cancer Center. Yuexiu District, Dongfeng East Road 651, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No